CLINICAL TRIAL: NCT02528396
Title: A Randomized, Monocentric, Double-blind, Multiple Daily Dose, Two-period, 14 Day Cross-over Trial to Investigate the Efficacy, Pharmacokinetics, Safety and Tolerability of Individualized Doses of BioChaperone Insulin Lispro in Comparison to Humalog® U-100 in Patients With Type 1 Diabetes Mellitus
Brief Title: To Investigate the Efficacy and Safety of Individualized Doses of BioChaperone Insulin Lispro in Comparison to Humalog® U-100 in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BC3-CT013
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BioChaperone insulin lispro (Experimental)
  Interventions: Drug: BioChaperone insulin lispro
- Humalog® (Active Comparator)
  Interventions: Drug: Humalog®

INTERVENTIONS:
Drug: BioChaperone insulin lispro — Injection at t0,or t+15 minutes or t-15minutes with test meal
  Arms: BioChaperone insulin lispro
Drug: Humalog® — Injection at t0,or t+15 minutes or t-15minutes with test meal
  Arms: Humalog®

SUMMARY:
This is a double-blind, randomised, controlled, two period crossover phase Ib trial using an individualized standard meal with a fixed nutrient ratio in subjects with type 1 diabetes mellitus to investigate postprandial blood glucose control with BioChaperone insulin lispro compared to Humalog®. The assessments will be conducted before and after a period of multiple daily dose administrations for 14 days. The meal tolerance test will be performed on day 1-3 and on day 14 of each period. Furthermore the study aims at investigating Post-prandial glucose (PPG) profiles with BioChaperone insulin lispro and Humalog® when injected at various injection meal intervals (-15min, 0 minutes, +15 minutes).

Each subject will be randomised to a sequence of two treatments, either BioChaperone insulin lispro-Humalog® or Humalog®-Biochaperone insulin lispro, and three different sequences of injection-meal intervals. A blinded to patient continuous monitoring of glucose (CGM) will be performed during the 14 day treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) ≥ 12 months
* Treated with multiple daily insulin injections (no pump users) ≥ 12 months
* Current total daily insulin treatment <1.2 (I)U/kg/day
* Body mass index (BMI) 18.5-28.0 kg/m² (both inclusive)
* HbA1c (N-(1-deoxy)-fructosyl-haemoglobin) ≤ 9.0% by local laboratory analysis
* Fasting C-peptide ≤ 0.30 nmol/L

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products
* Type 2 diabetes mellitus
* Patients using continuous subcutaneous insulin infusion (CSII)
* Previous participation in this trial. Participation is defined as randomised
* The receipt of any investigational product within 3 months prior to this trial
* Clinically significant abnormal haematology, biochemistry, lipids, or urinalysis screening tests, as judged by the Investigator considering the underlying disease
* Presence of clinically significant acute gastrointestinal symptoms (e.g. nausea, vomiting, heartburn or diarrhoea), as judged by the Investigator
* Known slowing of gastric emptying and or gastrointestinal surgery that in the opinion of the investigator might change gastrointestinal motility and food absorption
* Unusual meal habits and special diet requirements or unwillingness to eat the food provided in the trial

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
AUCΔBG0-2h (timepoint 0 = administration of the meal) | 2 hours
  Incremental area under the blood glucose (BG) concentration-time curve from 0-2 hours after a meal on day 1-3 [comparison between treatments Biochaperone insulin lispro vs. lispro (Humalog®)]
AUClispro 0-30min (timepoint 0 = time of dosing) | 30 minutes
  Area under the serum insulin lispro concentration-time curve from 0-30 minutes after bolus dose on one of days 1, 2 or 3 (comparison between treatments BioChaperone insulin lispro vs. lispro (Humalog®))

SECONDARY OUTCOMES:
AUClispro_0-6h | 6 Hours
  Area under the serum insulin lispro concentration-time curve from 0-6 hours after bolus dose
Cmax_lispro | up to 6 Hours
  Maximum serum insulin lispro concentration
Tmax_lispro | up to 6 Hours
  Time to maximum observed serum insulin lispro concentration
AUCBG_0-6h | 6 Hours
  Area under the curve under the blood glucose (BG) concentration time curve from 0-6 hours
ΔBGmax | 6 Hours
  Maximum blood glucose (BG) excursion after a standard meal (0-6 hours)
Adverse events | Up to 3 months
  Number of Adverse events
Local tolerability injection site reactions | 14 days
  Injection site reactions over 14 days of exposure

CONTACTS AND LOCATIONS:
Overall Officials: Grit Andersen, MD, Principal Investigator — Profil GmbH
Locations (1):
- Profil GmbH, Neuss, Germany